CLINICAL TRIAL: NCT04034667
Title: Clinical Study of CT and MR in Prediction of Driving Genes and Response in Patients With Lung Cancer
Brief Title: Study of CT and MR in the Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FSK003
Record Dates: First submitted 2019-07-17; First posted 2019-07-26 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer Squamous Cell; CT; Genes; Response; MRI
Keywords: Lung Cancer; Imaging features; Driving genes; Prediction; Therapy response
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Lung cancer is one of the leading causes of cancer-related deaths in China. Despite advances in systemic therapy and improvement nonsurvival rates for patients with advanced lung cancer, morbidity and mortality remain high.

Recently, many studies reported that patients with positive driving genes such as EGFR(epidermal growth factor receptor,EGFR), ALK(anaplastic lymphoma kinase,ALK), ROS1(c-ros oncogene 1 receptor,ROS1), BRAF (V-raf murine sarcoma viral oncogene homolog B1, BRAF)and so on have clearly targeted drugs, which bring survival benefits to patients. However, about half of patients still lack a clear driving gene target, which may have improved survival due to higher response rates to radiation therapy and other chemotherapy medications.

Development of noninvasive imaging biomarkers such as CT (computed tomography,CT)and MRI (magnetic resonance imaging,MRI)may not only evaluate the response to therapy ,but also could predict the efficacy of drug therapy and whether the driving gene is positive or not, through analysing the relationship between clinical related data and imaging features to find the imaging characteristics for making clinical decisions, and, consequently, contribute to an improved prognosis.

DETAILED DESCRIPTION:
To explore the value of CT and MR using multiple sequences, including T2-TSE-BLADE, T2 maps StarVIBE, and iShim-DWI in evaluating the driving genes and prediction of response to therapy and OS in patients with lung cancer.

Patients with biopsy-proven lung cancer were prospectively enrolled for imaging on CT and a 3T MRI scanner . The MRI protocol included T2-TSE-BLADE, T2 maps,iShim-DWI and StarVIBE sequences, and so on. Patients received treatment according to NCCN( National Comprehensive Cancer Network) guideline. CT and MRI features were analyzed to find the correlation between pretreatment imaging features and driving genes and therapy response. The study will include 400 patients. Inter-reader agreements of TN staging were analyzed excellent for CT and MRI. Diagnostic accuracy of CT and MRI will be calculated separately.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with preoperative pathologically con-firmed lung cancer by endoscopy and preoperative imaging data were included.
2. No contraindications for MRI examination. No contraindications for iodinated contrast.
3. The patients participate in this study with informed consent.

Exclusion Criteria:

1. The patients couldn't performed MSCT or MR scanning or artefacts affect the evaluation.
2. The patients are extremely anxious and uncooperative about surgery or neoadjuvant therapy .
3. PatientsThe patients refuse to participate in the project.
4. Other situations considered by investigators not meet the inclusion criteria.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with biopsy-proven lung cancer will receive treatment
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Study of relationship between clinical related data(driving genes and response) and imaging features(MSCT and MRI) in lung Cancer | up to 2 year
  Retrospectively reviewed data for patients diagnosed with lung cancer . All patients had received a histopathologic diagnosis of lung cancer based on bronchoscopic, percutaneous needle-guided, or surgical biopsies and had undergone gene mutation studies. Analysed the relationship between clinical related data(driving genes and response) and imaging features.
MSCT and MRI prediction of prognosis in lung cancer | up to 2 year
  To construct a model,a depth convolution neural network based on MSCT and multi-modal MR quantitative images which can automatically mine key images characterization, combined with imaging features,driving genes and prognosis,could further help to improve the prediction of response and OS of lung cancer treated with systematic therapy .

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shi L, Rong Y, Daly M, Dyer B, Benedict S, Qiu J, Yamamoto T. Cone-beam computed tomography-based delta-radiomics for early response assessment in radiotherapy for locally advanced lung cancer. Phys Med Biol. 2020 Jan 10;65(1):015009. doi: 10.1088/1361-6560/ab3247. PMID 31307024
- [Background] Lee G, Lee HY, Park H, Schiebler ML, van Beek EJR, Ohno Y, Seo JB, Leung A. Radiomics and its emerging role in lung cancer research, imaging biomarkers and clinical management: State of the art. Eur J Radiol. 2017 Jan;86:297-307. doi: 10.1016/j.ejrad.2016.09.005. Epub 2016 Sep 10. PMID 27638103
- [Background] Akinci D'Antonoli T, Farchione A, Lenkowicz J, Chiappetta M, Cicchetti G, Martino A, Ottavianelli A, Manfredi R, Margaritora S, Bonomo L, Valentini V, Larici AR. CT Radiomics Signature of Tumor and Peritumoral Lung Parenchyma to Predict Nonsmall Cell Lung Cancer Postsurgical Recurrence Risk. Acad Radiol. 2020 Apr;27(4):497-507. doi: 10.1016/j.acra.2019.05.019. Epub 2019 Jul 6. PMID 31285150
- [Background] Seki S, Fujisawa Y, Yui M, Kishida Y, Koyama H, Ohyu S, Sugihara N, Yoshikawa T, Ohno Y. Dynamic Contrast-enhanced Area-detector CT vs Dynamic Contrast-enhanced Perfusion MRI vs FDG-PET/CT: Comparison of Utility for Quantitative Therapeutic Outcome Prediction for NSCLC Patients Undergoing Chemoradiotherapy. Magn Reson Med Sci. 2020 Feb 10;19(1):29-39. doi: 10.2463/mrms.mp.2018-0158. Epub 2019 Mar 18. PMID 30880291
- [Background] Ciliberto M, Kishida Y, Seki S, Yoshikawa T, Ohno Y. Update of MR Imaging for Evaluation of Lung Cancer. Radiol Clin North Am. 2018 May;56(3):437-469. doi: 10.1016/j.rcl.2018.01.005. PMID 29622078